CLINICAL TRIAL: NCT06558916
Title: Comparison of the Analgesic Efficacy of Dexketoprofen Trometamol, Meperidine, and Paracetamol in Patients Presenting With Renal Colic
Brief Title: Comparison of the Analgesic Efficacy of Dexketoprofen Trometamol, Meperidine, and Paracetamol in Renal Colic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ismail Tekin (Other Government)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor-Investigator, Ismail Tekin, Principal Investigator, Primary Health Care Corporation, Qatar
Organization: Primary Health Care Corporation, Qatar (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ErciyesUniversity-IT01
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Analgesia; Renal Colic
Keywords: Analgesic efficacy; Dexketoprofen trometamol; Emergency department; Meperidine; Paracetamol; Renal colic
MeSH Terms: conditions — Agnosia; Renal Colic; Emergencies | interventions — dexketoprofen trometamol; Meperidine; Acetaminophen; Fentanyl

STUDY DESIGN:
Intervention Model Description: The patients were randomized and numbered using a computer. Ninety eligible patients diagnosed with renal colic and who agreed to participate in the study were included. Thirty patients were assigned to each of the three groups-dexketoprofen trometamol, meperidine and paracetamol.The study drugs were administered to patients suspected of having renal colic in random order: dexketoprofen trometamol IV 50 mg (ampoule containing Dexalgin 50 mg injectable solution), meperidine IV 50 mg (Aldolan 100 mg ampoule) and paracetamol IV 1000 mg (Perfalgan 10 mg/mL infusion solution) was prepared as a 250 mL solution in standard saline, with the same appearance. The drugs were given as a single dose over 15 minutes.
Who Masked: Participant, Care Provider
Masking Description: The physician who evaluated the patient ordered the analgesic X. Before the evaluation, the patients were informed about the pain scales to be used in the study, namely the visual analog scale (VAS) and verbal rating scale (VRS). The patients then made VAS and VRS markings on the evaluation forms without looking at the previous marking location. Neither the patients nor the physicians knew which study group they were in during the clinical practice phase, as the study was double-blind.
  The study drugs were administered to patients suspected of having renal colic in random order with the same appearance. The nurse who prepared the solution was informed about the study, but the nurse who administered the drug did not know which group the patient was in.
Oversight: FDA-regulated Drug: No

ARMS (3):
- Dexketoprofen trometamol (Experimental): The study drugs were administered to patients suspected of having renal colic in random order: dexketoprofen trometamol IV 50 mg (ampoule containing Dexalgin 50 mg injectable solution) was prepared as a 250 mL solution in standard saline, with the same appearance. The drugs were given as a single dose over 15 minutes.
  Interventions: Drug: Dexketoprofen Trometamol; Drug: Fentanyl
- Meperidine (Experimental): The study drugs were administered to patients suspected of having renal colic in random order: meperidine IV 50 mg (Aldolan 100 mg ampoule) was prepared as a 250 mL solution in standard saline, with the same appearance. The drugs were given as a single dose over 15 minutes.
  Interventions: Drug: Meperidine Injectable Solution; Drug: Fentanyl
- Paracetamol (Experimental): The study drugs were administered to patients suspected of having renal colic in random order: paracetamol IV 1000 mg (Perfalgan 10 mg/mL infusion solution) was prepared as a 250 mL solution in standard saline, with the same appearance.The drugs were given as a single dose over 15 minutes.
  Interventions: Drug: Paracetamol; Drug: Fentanyl

INTERVENTIONS:
Drug: Dexketoprofen Trometamol
  Other Names: Arveles; Dexalgin
  Arms: Dexketoprofen trometamol
Drug: Meperidine Injectable Solution
  Other Names: Pethidine; Aldolan
  Arms: Meperidine
Drug: Paracetamol
  Other Names: Acetaminophen; Parol
  Arms: Paracetamol
Drug: Fentanyl — Patients with a VAS score of 40 mm or higher at the 30th minute were given fentanyl (1 mcg/kg, intravenously) as a rescue drug.
  Other Names: Sublimaze

SUMMARY:
This study aimed to compare the effectiveness of intravenous (IV) dexketoprofen trometamol, IV meperidine, and IV paracetamol as analgesics for renal colic in patients at the Emergency Department of Erciyes University Medical School. The double-blind, randomized trial included 90 patients aged 18-65 years. Patients were divided into three groups of 30, receiving 50 mg IV dexketoprofen trometamol, 50 mg IV meperidine, or 1000 mg IV paracetamol, administered in 250 mL of saline over 15 minutes. Pain intensity was measured at 15, 30, and 60 minutes post-administration using a 100-mm visual analog scale (VAS) and a 4-point verbal rating scale (VRS). Successful treatment was defined as a 50% or greater reduction in VAS score at 30 minutes. Patients with a VAS score of 40 mm or higher at the 30th minute were given fentanyl (1 mcg/kg, intravenously) as a rescue drug.

DETAILED DESCRIPTION:
Study design

This clinical trial was conducted at a single center, involving a prospective, randomized, double-blind study. The main objective was to compare the analgesic effectiveness of three different medications-IV dexketoprofen trometamol, IV meperidine, and IV paracetamol in patients who arrived at the emergency department with renal colic.

Selection of participants

Patients who had taken any analgesic medication in the six hours preceding their arrival, those who had a regular medication schedule, individuals under 18 years of age or over 65, hemodynamically unstable patients, patients with renal, hepatic, cardiac, or respiratory failure, those allergic to the drugs used in the study, pregnant or breastfeeding women, those with a history of renal transplantation, patients with only one kidney, individuals with serum creatinine levels exceeding 2 mg/dL, those with a history of gastrointestinal bleeding and peptic ulcer, and patients unable to fill out the pain scale due to vision problems were excluded from the study.

The patients were randomized and numbered using a computer. Ninety eligible patients diagnosed with renal colic and who agreed to participate in the study were included. Thirty patients were assigned to each of the three groups-dexketoprofen trometamol, meperidine and paracetamol.

Interventions

All patients who presented to our emergency department with symptoms and signs indicative of renal colic were interviewed to gather information on their medical history. A detailed physical examination was then performed, and exclusion criteria were assessed. The patients were informed about the study and consent was obtained. Vascular access was established for all patients, and Complete Blood Count (CBC), Blood Urea Nitrogen (BUN) Creatinine, Sodium, Potassium and Aspartate aminotransferase (AST), Alanine transaminase (ALT), and urinalysis tests were requested for diagnosis and differential diagnosis. During the blood draw, the physician who evaluated the patient ordered the analgesic X. Before the evaluation, the patients were informed about the pain scales to be used in the study, namely the visual analog scale (VAS) and verbal rating scale (VRS). The patients then made VAS and VRS markings on the evaluation forms without looking at the previous marking location. Neither the patients nor the physicians knew which study group they were in during the clinical practice phase, as the study was double-blind.

The study drugs were administered to patients suspected of having renal colic in random order: dexketoprofen trometamol IV 50 mg (ampoule containing Dexalgin 50 mg injectable solution), meperidine IV 50 mg (Aldolan 100 mg ampoule) and paracetamol IV 1000 mg (Perfalgan 10 mg/mL infusion solution) was prepared as a 250 mL solution in standard saline, with the same appearance. The nurse who administered the drug was informed about the study, but the nurse who prepared the solution did not know which group the patient was in. The drugs were given as a single dose over 15 minutes.

Direct Urinary System X-ray and Urinary Ultrasound Sonography (USG) were conducted to detect stones and signs of urinary system obstruction in patients with renal colic. In cases where the diagnosis of renal colic was unclear, Computed Tomography was conducted for diagnosis and differential diagnosis. The study included 90 patients of both genders, aged between 18 and 65, who were diagnosed with renal colic after anamnesis, physical examination, laboratory and imaging tests, and who gave their consent to participate in the research. Statistical analyses were then performed.

If any unexpected effect was observed in the patients during the study period, the patient did not accept the treatment or wanted to leave the study; such patients were excluded from the study in the preparation phase. Fortunately, no such situation was encountered during the follow-ups.

Methods of measurements

The time at which treatment began was recorded as 0th minutes and pain levels were measured using the VAS scale, which ranges from "0 mm (no pain)" to "100 mm (unbearable pain)". The pain levels were measured before treatment and at the 15th, 30th and 60th minutes after the treatment. Pain severity was evaluated using VRS and classified as "none"-"mild"-"moderate"-"severe".

A treatment was considered successful if there was a 50% or greater reduction in the VAS score at the 30th minute [8]. If a patient's VAS score was ≥40 mm at the 30th minute, they were given 1 mcg/kg of Fentanyl IV as a rescue medication. All patients were monitored for at least 60 minutes, and any side effects and vital signs were recorded during this period.

Data analysis

Statistical analysis conducted in this study involved the use of various methods such as t-test independent samples, one-way variance analysis, and variance analysis in repeated measurements. The categorical variables were analyzed using the chi-square test. The numerical variables were expressed as arithmetic mean standard deviation (mean ± SD). Any p-value less than 0.05 was considered statistically significant. The statistical analysis was performed using version 22 of the "SPSS for Windows" package program (IBM, Armonk, NY, United States).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65.
* Diagnosed with renal colic via anamnesis, physical examination, laboratory, and imaging tests.
* Provided informed consent to participate in the research.
* Both genders.

Exclusion Criteria:

* Recent intake of any analgesic medication within six hours prior to arrival.
* Regular medication schedule.
* Age under 18 or over 65.
* Hemodynamically unstable patients.
* Renal, hepatic, cardiac, or respiratory failure.
* Allergies to study drugs.
* Pregnant or breastfeeding women.
* History of renal transplantation.
* Presence of only one kidney.
* Serum creatinine levels exceeding 2 mg/dL.
* History of gastrointestinal bleeding or peptic ulcer.
* Inability to complete the pain scale due to vision problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
VAS score change at the 30th minute | 0th minute and 30th minute
  The time at which treatment began was recorded as 0th minutes and pain levels were measured using the VAS scale, which ranges from "0 mm (no pain)" to "100 mm (unbearable pain)". The pain levels were measured before treatment and at the 15th, 30th and 60th minutes after the treatment. Pain severity was evaluated using VRS and classified as "none"-"mild"-"moderate"-"severe".
  A treatment was considered successful if there was a 50% or greater reduction in the VAS score at the 30th minute.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Tekin, Principal Investigator — Primary Health Care Corporation

IPD SHARING:
Plan to Share IPD: No